CLINICAL TRIAL: NCT00004433
Title: Randomized Study of Pergolide in Children With Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/13395; MUSC-6130; MUSC-FDR001111
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-03

CONDITIONS: Tourette Syndrome
Keywords: Tourette syndrome; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Tourette Syndrome; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Pergolide

INTERVENTIONS:
Drug: pergolide

SUMMARY:
OBJECTIVES:

I. Evaluate the presumed mechanism of action of low dose pergolide to act acutely through the dopaminergic autoreceptor or postsynaptically at D2 sites in children 7 to 17 with tourette syndrome (GTS).

II. Compare tolerability and safety of pergolide in these patients to standard neuroleptic therapy via naturalist assessment after 3-6 months of treatment using matched historical controls on neuroleptics.

III. Determine efficacy of pergolide for tic control in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a three part study: part I is a randomized, double blind, fixed single dose study; part II is a randomized, open label, stratified study; and part III is a randomized, double blind, placebo controlled study.

Part I patients are randomized to receive oral pergolide at one of three dose levels or placebo for 10 weeks. Part II patients are randomized to receive either low or high dose pergolide for 4 weeks.

Part III patients are randomized to first receive either pergolide or placebo by oral fixed doses twice daily followed by flexible clinically adjusted dosing for the next 3 weeks after a 2-week placebo run-in. Patients then cross over to receive the other treatment after another 2 weeks of placebo run-in. Total treatment duration is 16 weeks.

Patients are followed at 6 months.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

DSM IV primary diagnosis of Tourette syndrome (GTS) Multiple Axis I and Axis II diagnoses allowed

Tourette symptom severity great enough to warrant medication (CGI severity index at least 4)

No chronic motor tic disorder or transient tic disorder, anorexia nervosa, pervasive developmental disorders, substance/alcohol abuse or dependence within the past year, schizophrenia or any psychotic disorder

--Prior/Concurrent Therapy--

At least 4 weeks since prior neuroleptic therapy

At least 2 weeks since all other prior medications

No concurrent neuroleptic therapy or psychotropic therapy (i.e., antidepressant or anticholinergic)

No concurrent medication that may alter or interact with pergolide

--Patient Characteristics--

Performance status: Outpatient status

Hematopoietic: Normal or clinically insignificant values

Hepatic: Normal or clinically insignificant values

Renal: Normal or clinically insignificant values

Cardiovascular: Normal electrocardiogram

Other: No serious or unstable medical illness (i.e., diabetes, seizure disorder); Must be able to perform required measurements (i.e., no low I.Q.); Effective contraception required by all fertile patients

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74
Dates: Start 1994-12; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Floyd R. Sallee, Study Chair — Medical University of South Carolina

REFERENCES:
- [Background] Griesemer DA. Pergolide in the management of Tourette syndrome. J Child Neurol. 1997 Sep;12(6):402-3. No abstract available. PMID 9309526
- [Background] Lipinski JF, Sallee FR, Jackson C, Sethuraman G. Dopamine agonist treatment of Tourette disorder in children: results of an open-label trial of pergolide. Mov Disord. 1997 May;12(3):402-7. doi: 10.1002/mds.870120320. PMID 9159736